CLINICAL TRIAL: NCT03089216
Title: Combined Bleaching Technique: Efficacy and Tooth Sensitivity - A Randomized, Double Blind Clinical Trial
Brief Title: Combined Bleaching Technique: Efficacy and Tooth Sensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Terezinha de Jesus Esteves Barata (Other)
Responsible Party: Sponsor-Investigator, Terezinha de Jesus Esteves Barata, tde Jesus Esteves Barata, Universidade Federal de Goias
Organization: Universidade Federal de Goias (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 043178
Record Dates: First submitted 2017-03-17; First posted 2017-03-24 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Tooth Bleaching; Tooth Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Arginine; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combined Bleaching(2x20) (Experimental): In-office: 35% hydrogen peroxide of 20 minutes each. At-home: 10% carbamide peroxide
  Interventions: Procedure: Combined Bleaching(2x20)
- Combined Bleaching(2x20) with arginine (Experimental): Combined Bleaching(2x20) with arginine In-office: 35% hydrogen peroxide of 20 minutes each. At-home: 10% carbamide peroxide Desensitizing agent: dentifrice containing 8% arginine and calcium carbonate.
  Interventions: Procedure: Combined Bleaching(2x20) with arginine; Drug: 8% arginine and calcium carbonate
- Combined Bleaching(1x20) (Experimental): In-office: 35% hydrogen peroxide of 20 minutes each. At-home: 10% carbamide peroxide
  Interventions: Procedure: Combined Bleaching (1x20)
- Combined Bleaching(1x20) with arginine (Experimental): Combined Bleaching(1x20) with arginine In-office: 35% hydrogen peroxide of 20 minutes each. At-home: 10% carbamide peroxide Desensitizing agent: dentifrice containing 8% arginine and calcium carbonate.
  Interventions: Procedure: Combined Bleaching(1x20) with arginine; Drug: 8% arginine and calcium carbonate

INTERVENTIONS:
Procedure: Combined Bleaching(2x20) — one clinical session with two applications of 35% hydrogen peroxide of 20 minutes each. 10% carbamide peroxide for two hours daily over the course of two weeks.
  Arms: Combined Bleaching(2x20)
Procedure: Combined Bleaching(2x20) with arginine — one clinical session with two applications of 35% hydrogen peroxide of 20 minutes each. 10% carbamide peroxide for two hours daily over the course of two weeks.
  Arms: Combined Bleaching(2x20) with arginine
Procedure: Combined Bleaching (1x20) — one clinical session with one application of 35% hydrogen peroxide of 20 minutes each. 10% carbamide peroxide for two hours daily over the course of two weeks.
  Arms: Combined Bleaching(1x20)
Procedure: Combined Bleaching(1x20) with arginine — one clinical session with one application of 35% hydrogen peroxide of 20 minutes each. 10% carbamide peroxide for two hours daily over the course of two weeks.
  Arms: Combined Bleaching(1x20) with arginine
Drug: 8% arginine and calcium carbonate — using during all the treatment.
  Other Names: dentifrice containing carbonate arginine
  Arms: Combined Bleaching(1x20) with arginine; Combined Bleaching(2x20) with arginine

SUMMARY:
The aim of this clinical study is to evaluate the efficacy and dental sensitivity associated with Combined Bleaching Technique (in-office + at-home) varying in-office bleaching application under two different time protocols, and dentifrice containing arginine 8% and carbonate calcium use. One hundred eight participants who meet the study inclusion criteria will be selected. The desensitizing agent used will be a dentifrice containing 8% arginine and calcium carbonate. In each evaluation will be determined: tooth sensitivity and color. The data collected will be submitted to the factorial statistical analysis for evaluation of color and chi-square test for tooth sensitivity (α = 5%).

DETAILED DESCRIPTION:
This study will be conducted under the CONSORT recommendations. After approval by the Ethics Committee for Research duly registered, the trial will be conducted in the clinic of dental school at the Federal University of Goias located in Goiania. One hundred eight participants 108 volunteers will be selected on the criteria that qualify inclusion and exclusion from the study will be reported all volunteers were examined not qualify under the criteria for inclusion as part of the initial according to CONSORT recommendations .

After signing the signed an informed consent form all volunteer participants will receive a dental prophylaxis with pumice and water in a rubber cups for the removal of extrinsic stains two weeks before the beginning of tooth whitening.

ELIGIBILITY:
Inclusion Criteria:

* Upper and lower anterior teeth without restorations;
* Upper and lower anterior teeth that have never undergone a bleaching procedure and are A2 or darker in color compared to the Vita Classical).

Exclusion Criteria:

* Presence of primary and/or secondary carious lesion (s) on upper and lower anterior teeth;
* Presence of non-carious lesions, such as abfraction, erosion and abrasion;
* Presence of clinically visible cracks or defects of dental enamel on the dental surfaces of the upper and lower anterior teeth;
* Use of fixed orthodontic appliances;
* Presence of tooth sensitivity classified as equal to or greater than mild;
* Presence of severe dental dimming;
* Presence of parafunctional habits;
* Presence of any oral pathology;
* Smokers;
* pregnant and lactating women

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabella N Favarão, DDS, MS, Principal Investigator — Universidade Federal de Goias

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 325 participants were examined to check whether they met the inclusion and exclusion criteria; 217 participants were excluded because they presented initial conditions described in the exclusion criteria of the study; 108 were enrolled.
Groups:
- Combined Bleaching(2x20); Combined Bleaching(1x20): two 20-minute 35%HP applications (2x20); at-home bleaching was performed with 10% carbamide peroxide (CP) for two hours daily for 16 days.
- Combined Bleaching(1x20) With Arginine: one 20-minute 35%HP applications (2x20); at-home bleaching was performed with 10% carbamide peroxide (CP) for two hours daily for 16 days. dentifrice containing 8% arginine and calcium carbonate was used during all treatment.
- Combined Bleaching(2x20) With Arginine: two 20-minute 35%HP applications (2x20); at-home bleaching was performed with 10% carbamide peroxide (CP) for two hours daily for 16 days. dentifrice containing 8% arginine and calcium carbonate was used during all treatment.
Period: Overall Study
Arm/Group | Combined Bleaching(2x20) | Combined Bleaching(1x20) | Combined Bleaching(1x20) With Arginine | Combined Bleaching(2x20) With Arginine
Started | 27 | 27 | 27 | 27
Completed | 27 | 27 | 27 | 26
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Bleaching(2x20) | Combined Bleaching(1x20) | Combined Bleaching(1x20) With Arginine | Combined Bleaching(2x20) With Arginine | Total
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 27 | 27 | 108
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.8 (2.1) | 22.7 (3.1) | 20.7 (2.1) | 20.8 (1.7) | 21.2 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 17 | 21 | 69
  Male | 10 | 13 | 10 | 6 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Tooth Sensitivity (TS)
Description: Tooth sensitivity (TS) was evaluated using a five-point rating scale (NRS), in which 0 = none (minimum value), 1 = mild, 2 = moderate, 3 = considerable, and 4 = severe (maximum value); and a visual analogue scale (VAS) in wich each participant placed a line perpendicular to a 10-cm-long line (on which 0 referred to "no pain" (minimum value) and 10 referred to "severe pain" (maximum value)).
  Tooth sensitivity (TS) was evaluated during bleaching, and up to 48 hours postbleaching. The worst TS score or numeric value obtained in each assessment was considered for statistical purposes. It was calculated an average to obtain the median.
Time Frame: during bleaching, and up to 48 hours postbleaching
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Combined Bleaching(2x20) | Combined Bleaching(1x20) | Combined Bleaching(1x20) With Arginine | Combined Bleaching(2x20) With Arginine
Number analyzed (Participants) | 27 | 27 | 27 | 27
score on a scale
  Intensity of TS during bleaching (NRS scale) | 1 [0 to 1] | 1 [1 to 1] | 1 [0 to 1] | 0 [0 to 1]
  Intensity of TS up to 48 hours (NRS scale) | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Intensity of TS during bleaching (VAS scale) | 0.8 [0 to 8] | 0.9 [0 to 4] | 0.6 [0 to 6] | 0.3 [0 to 8]
  Intensity of TS up to 48 hours (VAS scale) | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 2] | 0 [0 to 0]

2. Secondary Outcome: Color Evaluation
Description: Objective color evaluation:
  The shade was determined using spectrophotometer VITA Easyshade, in which the parameters L*, a*, and b*, in which L* represents the value from 0 (black) to 100 (white) and a* and b* represent the shade, where a* is the measurement along the red-green axis and b* is the measurement along the yellow-blue axis.
  The color alteration (ΔE) was determined by the differences between the values obtained at baseline and one month after the treatment, which was calculated with the formula: ΔE = [(ΔL *) 2 + (Δa *) 2 + (Δb *) 2]1/2.
  In the Outcome Measure Data Table it was presented Mean and Standard Deviation of the color alteration (ΔE) between Baseline vs one month after bleaching for each group.
Time Frame: The evaluations were performed in the baseline period and one month after the treatment
Measure: Mean (Standard Deviation); unit: percentage of color change
Arm/Group | Combined Bleaching(2x20) | Combined Bleaching(2x20) With Arginine | Combined Bleaching(1x20) | Combined Bleaching(1x20) With Arginine
Number analyzed (Participants) | 27 | 26 | 27 | 26
percentage of color change | 8.28 (2.73) | 8.18 (2.76) | 7.72 (2.61) | 8.11 (2.76)

ADVERSE EVENTS:
Time Frame: Tooth sensitivity was evaluated at baseline and up to 48 hours after the combined bleaching.
Description: A five-point rating scale (NRS), in wich 0 = none, 1 = mild, 2 = moderate, 3 = considerable, and 4 = severe, as well as a visual analogue scale (VAS) was used to performed tooth sensitivity. Each participant placed a line perpendicular to a 10-cm-long line (on which 0 referred to "no pain" and 10 referred to "severe pain").
Arm/Group | Combined Bleaching(2x20) | Combined Bleaching(2x20) With Arginine | Combined Bleaching(1x20) | Combined Bleaching(1x20) With Arginine
Serious Adverse Events (participants affected / at risk) | 22/27 | 16/27 | 23/27 | 16/27
Other Adverse Events (participants affected / at risk) | 22/27 | 16/27 | 23/27 | 18/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Bleaching(2x20) (N=27) | Combined Bleaching(2x20) With Arginine (N=27) | Combined Bleaching(1x20) (N=27) | Combined Bleaching(1x20) With Arginine (N=27)
Tooth Sensitivity (Score of >3) (Investigations) | 22 (27) | 16 (27) | 23 (27) | 16 (27)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Bleaching(2x20) (N=27) | Combined Bleaching(2x20) With Arginine (N=27) | Combined Bleaching(1x20) (N=27) | Combined Bleaching(1x20) With Arginine (N=27)
Tooth Sensitivity (Score of <3) (Investigations) | 22 | 16 | 23 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT03089216/Prot_SAP_000.pdf